CLINICAL TRIAL: NCT07376707
Title: A Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics, and Antitumor Activity of TGI-5 as Monotherapy and in Combination With Nivolumab in Subjects With Locally Advanced/Metastatic Solid Tumors
Brief Title: A Phase 1 Study of TGI-5 as Monotherapy and in Combination With Nivolumab in Subjects With Locally Advanced/Metastatic Solid Tumors
Acronym: TGI5
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hefei TG ImmunoPharma Co., Ltd. (Other)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGI5-T1-01
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: CRC (Colorectal Cancer); Melanoma (Skin Cancer); HCC - Hepatocellular Carcinoma; NSCLC (Non-small Cell Lung Cancer)
Keywords: TGI-5; Locally Advanced/Metastatic Solid Tumors
MeSH Terms: conditions — Colorectal Neoplasms; Melanoma; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: In Phase 1a, subjects with histologically or cytologically diagnosed unresectable locally advanced/metastatic solid tumors.
  After screening, qualified subjects will be assigned to each cohort on a chronological basis. Subjects will receive TGI-5 at the assigned dose regimen (intravenous [IV] infusion), and the dose limiting toxicity (DLT) assessment will be conducted in the subjects during the DLT evaluation period (28 days after the first dose [i.e., Cycle 1, Day 1~Day 28]).
  In Phase 1b dose escalation part, subjects with histologically or cytologically diagnosed unresectable locally advanced/metastatic solid tumors.
  After screening, qualified subjects will be assigned to each cohort on a chronological basis. Subjects will receive TGI-5 at the assigned dose regimen in combination with a fixed dose of Nivolumab (240 mg, IV infusion) Q2W, and the DLT assessment will be conducted in the subjects during the DLT evaluation period (Cycle 1).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation of TGI-5 as monotherapy，Dose Escalation of TGI-5 in Combination with Nivolumab (Experimental): At the Phase 1a of this study, 0.01 mg/kg is proposed as the starting dose of TGI-5 as monotherapy for the FIH study. An accelerate titration and then traditional "3+3" dose escalation design will be used to explore the maximum tolerated dose (MTD)/optimal biological dose (OBD).
  Subjects will receive TGI-5 at the assigned dose regimen in combination with a fixed dose of Nivolumab (240 mg, IV infusion) Q2W, and the DLT assessment will be conducted in the subjects during the DLT evaluation period (Cycle 1).
  Interventions: Drug: TGI-5

INTERVENTIONS:
Drug: TGI-5 — Subjects will receive TGI-5 as monotherapy in Phase 1a by Q2W for 28-day cycles.
  Subjects will receive TGI-5 in combination with Nivolumab in Phase 1b by Q2W for 28-day cycles.
  Other Names: Nivolumab

SUMMARY:
This is a Phase 1, multicenter, open-label, two-parts, FIH study to evaluate the tolerability, safety, PK/PD, and preliminary antitumor activity of TGI-5 as monotherapy and in combination with Nivolumab in subjects with unresectable locally advanced/metastatic solid tumors.

The study consists of two parts: TGI-5 monotherapy (Phase 1a: including a dose escalation part and a dose expansion part), TGI-5 in combination with a fixed dose of Nivolumab (Phase 1b: including a dose escalation part and a dose expansion part).

DETAILED DESCRIPTION:
In Phase 1a, subjects with histologically or cytologically diagnosed unresectable locally advanced/metastatic solid tumors, mainly but not limited to CRC, hepatocellular carcinoma (HCC), melanoma, and NSCLC who have progressed despite all standard therapy or are intolerant of all standard therapy, or for whom no effective standard therapy exists will be enrolled.

After screening, qualified subjects will be assigned to each cohort on a chronological basis. Subjects will receive TGI-5 at the assigned dose regimen (intravenous [IV] infusion), and the dose limiting toxicity (DLT) assessment will be conducted in the subjects during the DLT evaluation period (28 days after the first dose [i.e., Cycle 1, Day 1~Day 28]). Subjects who experience a DLT will permanently discontinue the study treatment and be closely monitored until the toxicity has resolved to Grade 1 or baseline or as long as the investigator considers it stable and unsolvable. After 28-day of DLT evaluation period, subjects who did not experience a DLT will continue to receive TGI-5 as monotherapy at the same dose level once every 2 weeks (Q2W) until discontinuation of treatment for any reason, such as confirmed progressive disease, unacceptable toxicity, initiation of a new anticancer therapy, death, lost follow-up, withdrawal of informed consent, or at the discretion of the investigator due to safety or compliance, whichever occurs first.

At the Phase 1a of this study, 0.01 mg/kg is proposed as the starting dose of TGI-5 as monotherapy for the FIH study. An accelerate titration and then traditional "3+3" dose escalation design will be used to explore the maximum tolerated dose (MTD)/optimal biological dose (OBD).

After the OBD is determined by the safety monitoring committee (SMC), the corresponding cohort will be expanded at the OBD dose level for further assessment of safety, PK/PD, and antitumor activity. About 10~20 subjects with histologically or cytologically diagnosed unresectable locally advanced/metastatic solid tumors, mainly but not limited to CRC, HCC, melanoma, and NSCLC who have progressed despite all standard therapy or are intolerant of all standard therapy, or for whom no effective standard therapy exists will be enrolled.

After the primary analysis of Phase 1a, the SMC will discuss and decide whether the study can proceed to Phase 1b based on data available from Phase 1a. The proposed starting dose of TGI-5 in combination with Nivolumab will be at least 2 dose levels below the MTD/OBD identified for TGI-5 as a single agent in Phase 1a. The starting dose of TGI-5 in combination with Nivolumab will be selected by the SMC based on the available safety, tolerability, PK/PD, and antitumor activity data from the previous monotherapy phase (Phase 1a), non-clinical studies of combined administration will also be considered comprehensively.

The dose of Nivolumab is selected as fixed dose (240 mg) Q2W, which is consistent with the dosing interval of TGI-5.

The "3+3" design and definition of MTD are the same as that in Phase 1a. Definition of recommended phase 2 dose (RP2D) is the same as OBD in Phase 1a.

In Phase 1b dose escalation part, subjects with histologically or cytologically diagnosed unresectable locally advanced/metastatic solid tumors, mainly but not limited to CRC, HCC, melanoma, and NSCLC who have progressed despite all standard therapy or are intolerant of all standard therapy, or for whom no effective standard therapy exists will be enrolled.

After screening, qualified subjects will be assigned to each cohort on a chronological basis. Subjects will receive TGI-5 at the assigned dose regimen in combination with a fixed dose of Nivolumab (240 mg, IV infusion) Q2W, and the DLT assessment will be conducted in the subjects during the DLT evaluation period (Cycle 1). When TGI-5 and Nivolumab are administered on the same day, it is recommended that TGI-5 be administered first. After 28-day of DLT evaluation period, subjects who did not experience a DLT will continue to receive the combination regimen until discontinuation of treatment for any reason, such as confirmed progressive disease, unacceptable toxicity, initiation of a new anticancer therapy, death, lost follow-up, withdrawal of informed consent, or at the discretion of the investigator due to safety or compliance, whichever occurs first.

Treatment cycles will occur consecutively without interruption unless an AE leading to treatment interruption occurs. Subjects who experience a DLT will permanently discontinue study treatment (both TGI-5 and Nivolumab) and be closely monitored until the toxicity has resolved to Grade 1 or baseline or if the investigator considers it stable and unsolvable.

Once the MTD and/or RP2D of TGI-5 in combination regimen is identified and the safety profile has been reviewed by the SMC and is considered safe and tolerable for subjects based on the available data, the dose expansion part of Phase 1b in the study will start.

Subjects who meet eligibility criteria are planned to be enrolled into 4 cohorts based on their tumor types to evaluate the efficacy and safety of TGI-5 in combination with Nivolumab. At least 2 dosages will be evaluated and compared in each cohort of dose expansion part to identify an optimal dosage as the RP2D.

The dose expansion phase will consist of 4 cohorts tentatively designated as:

* Cohort 1: Unresectable locally advanced/metastatic CRC
* Cohort 2: Unresectable locally advanced/metastatic melanoma
* Cohort 3: Unresectable locally advanced/metastatic NSCLC
* Cohort 4: Other Unresectable locally advanced/metastatic solid tumors

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female subject age ≥18 years at the time of informed consent. 2. Phase 1a and dose escalation part of Phase 1b: Subjects with histologically or cytologically diagnosed unresectable locally advanced/metastatic solid tumors, mainly but not limited to CRC, HCC, melanoma, NSCLC.

Dose expansion part of Phase 1b:

* Cohort 1: Subjects with histologically or cytologically diagnosed unresectable locally advanced and/or metastatic CRC.
* Cohort 2: Subjects with histologically or cytologically diagnosed unresectable locally advanced and/or metastatic melanoma.
* Cohort 3: Subjects with histologically or cytologically diagnosed unresectable locally advanced and/or metastatic NSCLC.
* Cohort 4: Subjects with other histologically or cytologically diagnosed unresectable locally advanced/metastatic solid tumors.

  3. Subjects should have documented progression of disease despite all standard therapy or are intolerant of all standard therapy, or for whom no effective standard therapy exists. (Standard therapies are defined as treatments recommended by local guidelines, including but not limited to, chemotherapy, radiation, target therapies based on mutation status, immunotherapy, and surgery in general).

Dose expansion part of Phase 1b:

* Cohort 1: Subjects with unresectable locally advanced and/or metastatic CRC o At least 2 prior standard chemotherapy/therapy regimens are required with documented progression or intolerability to the treatment.

  * Standard chemotherapy regimens include all the following ones (if eligible and no contraindication): Fluoropyrimidine-containing regimen, and/or oxaliplatin-containing regimen, and/or irinotecan-containing regimen (treatment with a FOLFIRINOX regimen will count as 2 regimens).
  * With or without an anti-VEGF therapy (e.g., bevacizumab).
  * At least one of the anti-EGFR monoclonal antibodies (cetuximab or panitumumab) for KRAS wild-type subjects if clinically indicated.
  * For subjects with a known microsatellite instability high (MSI-H):

    1. Prior treatment with an at least 2 doses of approved or investigational immune checkpoint inhibitor is required with documented progression or intolerability to the treatment.
    2. Demonstrated disease progression after immune checkpoint inhibitor treatment as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (Appendix 5). The initial evidence of disease progression is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented disease progression, in the absence of rapid clinical progression. Once disease progression is confirmed, the initial date of disease progression documentation will be considered the date of disease progression.
    3. Progressive disease that has been documented within 12 weeks from the last dose of immune checkpoint inhibitor.

       Note: a line of therapy is generally considered >2 cycles of exposure to the same regimen followed by radiographically documented progression. Agents that are mechanistically similar (e.g., 5-fluorouracil and capecitabine) and are used interchangeably due to tolerability but not progression may be considered as components of the same regimen upon discussion with the medical monitor.
  * Subjects must have progressed while receiving or after of the last administration of their last line of standard therapy or be unable to tolerate any of these standard treatments.
  * Subjects who progressed on/within 3 months of adjuvant therapy with anti-PD-1 antibody will be allowed; subjects who received adjuvant chemotherapy and had recurrence/progression with development of unresectable or metastatic disease during or within 6 months of completion of the adjuvant chemotherapy can count this as a line of therapy.
* Cohort 2: Subjects with anti-PD-(L)1 antibody PD-1 relapsed/refractory melanoma

  * PD-1 refractory disease as defined as progression on treatment with anti-PD-1 antibody administered either as monotherapy or in combination with other checkpoint inhibitors (anti-CTLA4 antibody or anti-LAG-3 antibody) or other therapies. Anti-PD-1 treatment progression is defined by meeting all of the following criteria:

    1) Has received at least 2 doses of an approved or investigational anti-PD-1 antibody with documented progression or intolerability to the treatment.

    2) Demonstrated disease progression after anti-PD-1 treatment as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (Appendix 5). The initial evidence of disease progression is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented disease progression, in the absence of rapid clinical progression. Once disease progression is confirmed, the initial date of disease progression documentation will be considered the date of disease progression.

    3) Progressive disease that has been documented within 12 weeks from the last dose of anti-PD-1 antibody.
  * Subjects who progressed on/within 3 months of adjuvant therapy with anti-PD-1 antibody will be allowed; an adjuvant therapy will count as 1 prior line of therapy if received within the prior 6 months.
  * For patients with BRAF V600 mutations, treatment with BRAF and MEK inhibitors prior to initiation on trial is required, unless patients are intolerant of BRAF targeted therapy.
  * Treatment must have been discontinued for disease progression or intolerance to therapy.
* Cohort 3: Subjects with anti-PD-(L)1 antibody relapsed/refractory NSCLC

  o Anti-PD-(L)1 antibody refractory disease as defined as progression on treatment with anti-PD-(L)1 inhibitor administered either as monotherapy or in combination with platinum-based chemotherapy or other therapies. Anti PD (L)1 treatment progression is defined by meeting all of the following criteria:
  1. Has received at least 2 doses of an approved or investigational anti-PD-(L)1 inhibitor with documented progression or intolerability to the treatment.
  2. Has demonstrated disease progression after anti-PD-(L)1 inhibitor as defined by RECIST v1.1 (Appendix 5). The initial evidence of disease progression is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented disease progression, in the absence of rapid clinical progression. Once disease progression is confirmed, the initial date of disease progression documentation will be considered the date of disease progression.
  3. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-(L)1 inhibitor.

     o Subjects who progressed on/within 3 months of adjuvant therapy with anti PD (L)1 inhibitor will be allowed; an adjuvant therapy will count as 1 prior line of therapy if received within the prior 6 months.

     o Documented disease progression during or after platinum-based chemotherapy alone or intolerability to the treatment for subjects with contraindications to anti PD (L)1 inhibitors.
     * Patients with NSCLC with known oncogenic driver (including but not limited to EGFR, ALK, ROS, MET alterations) must have received and progressed past driver-specific therapy.
     * Treatment must have been discontinued for disease progression or intolerance to therapy.
* Cohort 4: Subjects with other histologically or cytologically diagnosed unresectable locally advanced/metastatic solid tumors All subject in Phase 1b must meet PD-L1 expression ≥1%. 4. Subjects must have at least one evaluable lesion in Phase 1a or at least one measurable lesion in Phase 1b as defined by RECIST v1.1 (Appendix 5) which has not received radiotherapy (or progressive disease after radiotherapy).

  5. ECOG PS (Appendix 6) of 0~2. 6. Life expectancy ≥3 months. 7. Subjects have sufficient baseline organ function and laboratory data meet the following criteria at enrollment:
* Hematological (without need for hematopoietic growth factor or transfusion support within 2 weeks prior to enrollment):

  1) ANC ≥1.5×109/L. 2) Hemoglobin (HGB) ≥90 g/L. 3) Platelet (PLT) ≥75×109/L.
* Hepatic:

  1) AST and ALT ≤2.5×ULN (≤5×ULN for subjects with liver metastases). 2) Total bilirubin (TBil) ≤1.5×ULN, or TBil ≤3.0×ULN for subjects with liver cancer or liver metastases. Subjects with Gilbert's syndrome may enroll if direct bilirubin ≤1.5×ULN.
* Renal:

  1) Creatinine apparent clearance (CL) >50 mL/min according to modification Cockcroft-Gault equation (140-age [year])×body weight [kg]×1.23×(0.85 if female)/serum creatinine [μmol/L]).
* Coagulation:

  1) International normalized ratio (INR) ≤1.5. 2) Activated partial thromboplastin time (APTT) ≤1.5×ULN. 8. Woman of child-bearing potential must have a negative serum pregnancy test within 7 days prior to treatment. A female subject of nonchildbearing potential will have had at least 12 continuous months of natural (spontaneous) amenorrhea, follicle stimulating hormone level ≥40 mIU/mL at screening, and an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms), or have had surgical bilateral oophorectomy, hysterectomy, or tubal ligation ≥6 weeks prior to screening.

  9. Female subjects of childbearing potential or male subjects with a partner of childbearing potential must agree to use effective contraception at the time of informed consent and continuing through the study until 6 months after the last dose of study treatment (Appendix 4).

Exclusion Criteria:

* 1. Subject with known active central nervous system (CNS) primary tumor or metastases.

Note: Subject with previously treated CNS primary tumor/metastases can participate provided they are clinically stable for at least 2 weeks, have no evidence of new or enlarging brain metastases, and there has been no increase in steroid dose for 14 days prior to the first dose of TGI-5 to manage CNS symptoms. Subjects with carcinomatous meningitis or leptomeningeal spread, or spinal cord compression are excluded regardless of clinical stability.

2. History of intercurrent severe chronic or active infections:

1. Subjects with active hepatitis B, defined as: if hepatitis B virus surface antigen (HbsAg) positive, hepatitis B virus (HBV) deoxyribonucleic acid (DNA) assay should be performed, and HBV DNA is above the limit quantification.
2. Subjects with active hepatitis C, defined as: if hepatitis C virus (HCV) antibody positive, HCV ribonucleic acid (RNA) assay should be performed, and HCV RNA is positive.
3. Known history of acquired immune deficient syndrome (AIDS) or human immunodeficiency virus (HIV) infection.
4. Subjects with HIV infection may be eligible if CD4+ T cell counts ≥350 cells/µL and without a history of AIDS-defining opportunistic infections.
5. Other severe chronic within 4 weeks prior to the first dose of TGI-5, including but not limited to hospitalization for complications of infection, bacteremia, severe pneumonia, or active tuberculosis. Or uncontrolled active infections or unexplained fever >38°C within 7 days prior to first dose of TGI-5.

3. Has a history of active autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior the first dose of study drug.

With the following exceptions: clinically stable autoimmune thyroid disease; treatment with inhaled or topical corticosteroids such as ocular, intra-articular, and intranasal ≤10 mg daily of prednisone equivalent; short-term use of corticosteroids (no more than 7 days) for prophylaxis (e.g., to prevent contrast medium allergy or non-autoimmune allergic diseases); and replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes, physiologic corticosteroid replacement for adrenal or pituitary insufficiency).

4. Has a history of symptomatic interstitial lung disease. 5. Toxicities of prior therapies have not been resolved to Grade ≤1 or baseline as per NCI-CTCAE v5.0, except for alopecia, skin hyperpigmentation, Grade 2 neuropathy and Grade 2 endocrinopathy that is well controlled by replacement therapy.

6. Subjects with severe or uncontrolled cardiovascular disorder requiring treatment, including any of the following:

1. New York Heart Association (NYHA) class III or IV congestive heart failure.
2. Left ventricular ejection fraction (LVEF) <50% assessed by multiple-gated acquisition (MUGA) scan or echocardiogram (ECHO).
3. Mean ECG QT interval corrected by Fridericia's formula (QTcF) >480 milliseconds (ms) obtained from triplicate 12-lead ECGs, or congenital long QT syndrome.
4. Any of the following within 6 months prior to screening: Grade >2 ventricular arrhythmia, myocardial infarction, severe/unstable angina (even if controlled with medication), coronary artery bypass graft, congestive heart failure, cerebrovascular accident, or transient ischemic attack.
5. Presence of uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg). Subjects with a history of hypertension are allowed if blood pressure is controlled to within these limits by anti-hypertensive treatment.
6. Symptomatic pulmonary embolism within 6 months prior to initiation of study treatment.

7. Prior allogenic or autologous bone marrow transplantation or other solid organ transplantation.

8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years (Note: Subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and localized prostate cancer who have undergone potentially curative therapy. These subjects are not excluded).

9. Evidence of clinically significant immunosuppression such as the following:

1. Primary immunodeficiency state such as severe combined immunodeficiency disease (SCID).
2. Concurrent opportunistic infection. 10. Presence of uncontrolled pleural effusion, pericardial effusion or ascites requiring recurrent drainage procedures (monthly or more frequently).

11. Previously treated with the following antitumor therapy (prior to the first dose of TGI-5):

1) Previous treated with TIGIT-targeting therapy. 2) Chemotherapy, target therapy, immunotherapy, or other anticancer therapy within 28 days or 5 half-lives, whichever is shorter, prior to the first dose of study treatment, except:

1. Washout period for nitrosoureas or mitomycin is ≤6 weeks.
2. ≤5 half-lives or 2 weeks (whichever is longer) for fluoropyrimidines or small-molecule targeted agents.
3. Washout period for herbal therapy with anticancer indications is ≤2 weeks.
4. Anti-PD-1/PD-L1 antibody therapy within 6 weeks. 3) Prior radiotherapy ≤4 weeks prior to the first dose of study treatment, with the exception of a single fraction of radiotherapy for the purposes of palliation, which is permitted.

   4) Subject participated in any other clinical study and has received an investigational product within 28 days prior to the first dose of TGI-5.

   12. Has received systematic immunomodulatory drugs within 14 days before the first dose of study drug, such as thymosin, IL-2, and IFN.

   13. Has received a live vaccine within 4 weeks prior to the first dose of study drug.

   14. Has a recent major surgery within 4 weeks prior to the first dose of study drug or is expected to undergo major surgery during the study.

   15. Subject requiring anticoagulant treatment which cannot be safely interrupted, if medically needed for a study procedure (e.g., biopsy) based on the opinion of the investigator.

   16. Subjects who have experienced Grade ≥3 irAEs from prior immunotherapies or who discontinue immunotherapy due to immune-related toxicities.

   Note: Subjects with stable hypothyroidism on hormone replacement therapy are eligible.

   17. Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.

   18. Pregnancy or lactation. Women who are willing to discontinue breastfeeding prior to administration of study drug and do not intend to resume breastfeeding may be enrolled.

   19. Has known hypersensitivity to either the drug substances or inactive ingredients in the drug product.

   20. Pre-existing other serious medical conditions (e.g., active or chronic inflammatory lung disease have not resolved, uncontrolled acute or chronic nephropathy, uncontrolled pancreatitis, uncontrolled hepatopathy, uncontrolled diabetes mellitus, active gastric ulcer, gastrointestinal hemorrhage, uncontrolled epileptic seizure, and signs and symptoms of severe coagulopathy), familial or endemic disease that, in the opinion of the investigator, will interfere with planned staging, treatment, and follow-up, subject compliance, or will place the subject at high risk for treatment-related complications.

   21. Subjects who are unwilling or unable to comply with study procedures and study restrictions, or in the judgment of the investigator, would make the subject inappropriate for entry into this study.

   22. Subjects who have contraindication for use of PD-1/PD-L1 antibody (only for Phase 1b).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | First 28 days of treatment.
  The incidence of DLTs during the DLT assessment period
Frequency and Severity of Adverse Events (AE) | Screening to 30 days from last dose
  The incidences and percentages of patients experiencing AEs summarized by NCI CTCAE version 5.0 grade and by causality.

SECONDARY OUTCOMES:
Pharmacokinetics of TGI-5 | Day 1 of dosing through 30 days post last dose
  Maximum Plasma Concentration (Cmax)
Objective Response Rate (ORR) | Approximately 2 years.
  ORR according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, Doctorate, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The clinical trial has not yet been completed, and the relevant test results have not been statistically analyzed. Furthermore, this is classified business information and will not be made public for the time being.